CLINICAL TRIAL: NCT06166329
Title: Interest of the Chair Lift Test in the Prognostic Evaluation of Pulmonary Embolism: a Single-center Open Prospective Study
Acronym: SIT-EP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/0386/HP
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Non-severe Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chair lift test (Experimental)
  Interventions: Other: chair lift test

INTERVENTIONS:
Other: chair lift test — repetitions of the sit-stand position at a self-timed speed (safe and comfortable) as many times as possible for 1 minute

SUMMARY:
The objective of the study is to evaluate the prognostic performance of the chair lift test in the initial assessment of the severity of non-severe pulmonary embolism in hospitalized patients, in comparison with the current pulmonary embolism risk stratification score using the sPESI score refined by the use of cardiac biomarkers and right ventricular dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary embolism according to clinical algorithm, confirmed by thoracic angioscan or ventilation perfusion (V/P) scan,
* Non-serious pulmonary embolism, not requiring intensive care (thrombectomy or fibrinolysis not considered).
* sPESI score ≥ 1 [or = 0 with elevated troponin or presence of markers of VD dysfunction, or = 0 with need for hospitalization due to comorbidities unrelated to PE (social isolation, comprehension disorders, intercurrent infection, chronic renal failure, advanced cancer...)
* Patients with no contraindications to chair lift testing (no O2 at the time of testing).
* Effective anticoagulation for at least 1 hour.

Exclusion Criteria:

* sPESI score = 0 with outpatient referral.
* Diagnostic confirmation of Pulmonia Embolism by thoracic angioscan or scintigraphy more than 24h after suspicion of diagnosis.
* Hospitalization > 24h after introduction of anticoagulation, with subsequent confirmation by scintigraphy.
* Any sign of serious Pulmonia Embolism, requiring hospitalization in an intensive care unit.
* Asymptomatic Pulmonia Embolism discovered by chance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the one-minute chair rise test in comparison with the gold standard refined by the use of cardiac biomarkers and right ventricular dysfunction | 1 day

SECONDARY OUTCOMES:
Troponin measurement | 1 day
Presence or absence of post-pulmonary embolism dyspnea | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Delphine SIMON, MD, Principal Investigator — University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No